CLINICAL TRIAL: NCT04870294
Title: PBS CIMMO DTA® Cement in Post-operative Sensitivity: Randomized Clinical Trial
Brief Title: Dental Cement in Post-operative Sensitivity: Randomized Clinical Trial
Acronym: Bioactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, José Dias da Silva Neto, Professor Doctor, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Clinical study
Record Dates: First submitted 2021-03-07; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Restored Decayed Teeth and Post-operative Sensitivity
Keywords: Dentistry, Operative; Dental Restoration, Permanent; Dental Caries; Dental Pulp Capping; Dental Materials
MeSH Terms: conditions — Dental Caries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Comparison of two types of intervention: composite resin restoration and cavity lining before composite resin restoration.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study has double blind masking: as for patients and professional evaluator of the results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teeth treated with composite resin, control group (Active Comparator): The teeth grouped in group R were treated with composite resin restoration without liner material, considered a control group.
  Interventions: Device: Teeth treated with composite resin, control group
- Teeth treated with lining, pulp wall with PBS DTA® cement and composite resin restoration (Experimental): The teeth grouped in group D received PBS CIMMO DTA® as indirect capping material of the cavity, followed by restoration of composite resin.
  Interventions: Device: Teeth treated with lining, pulp wall with PBS DTA® cement and composite resin restoration

INTERVENTIONS:
Device: Teeth treated with composite resin, control group — The teeth grouped in group R were treated with composite resin restoration without liner material.
  Other Names: Filtek Z350 XT® composite resin (3M ESPE Dental Products TM, St. Paul, MN, USA)
  Arms: Teeth treated with composite resin, control group
Device: Teeth treated with lining, pulp wall with PBS DTA® cement and composite resin restoration — The teeth grouped in group D received PBS CIMMO DTA® as indirect capping material of the cavity, followed by restoration of composite resin.
  Other Names: PBS CIMMO DTA® cement.
  Arms: Teeth treated with lining, pulp wall with PBS DTA® cement and composite resin restoration

SUMMARY:
Context: CEMENT PBS CIMMO DTA® has physical and biological properties that classify it as a biocompatible material and inducer of biomineralization, attributes that qualify it as material as an indirect pulp capper in permanent tooth restorations. Objective: The present clinical study proposes the use of PBS CIMMO DTA® cement as an indirect pulp capper, in resin restorations composed of permanent molars and premolars. The objective was to minimize postoperative sensitivity arising from restorative procedures. Method: Randomized clinical trial with two arms, double blind, interventional, prospective. The sample consisted of 20 male patients, with an average age of 20 years. Totaling 70 teeth to be treated. The teeth were divided into two groups: Group R (Control Group, n = 35), treated with a standard restorative procedure. Group D (Study group n = 35), treated using CEMENT PBS CIMMO DTA®, as an indirect capper of the pulp wall. The evaluation was carried out by a masked examiner for both groups. Sensitivity tests were performed before the restorative procedure, at 48 hours, 7, 15 and 30 days after the procedure. The analysis included pain caused by thermal stimuli: Cold Test (TM); horizontal (TPH) and vertical (TPV) percussion; Bite Test (TM) and Pain Decline Time (DD) was measured. Measured using Visual Analog Scale (EVA).

DETAILED DESCRIPTION:
The present study is a clinical trial: an intervention model, prospective, randomized, double-blind (patients and evaluator). It was held at the Dental Office of the 14th Field Artillery Group - Pouso Alegre (MG), Military Organization of the Brazilian Army in conjunction with the University of Vale do Sapucaí (UNIVÁS), Pouso Alegre, Minas Gerais, Brazil; in the period from 23 March 2020 to 18 January 2021.

Participants were initially evaluated according to the inclusion and non-inclusion criteria of the research. Clinical examinations were performed initially using a mouth mirror, explorer probe (Golgran®, São Caetano do Sul, SP, Brazil). The data were recorded on clinical records for screening. The radiographic examination included performing periapical radiographs as diagnostic aids, for participants who met the inclusion criteria during the clinical examination. Oral hygiene guidelines were provided to all research participants. To begin the service, an anamnesis form was filled out.

Randomization occurred after applying the inclusion and non-inclusion criteria of the patients, 20 were selected, according to the initial clinical examination.

The 20 patients were randomized and the random sequence for submission to radiographic examinations was determined, defining 70 teeth to be treated, within the study criteria.

As for the group that each tooth would belong to; 70 brown envelopes were made: 35 containing green paper, belonging to the standard restorative procedure group and 35 containing pink paper, belonging to the DTA® group. Before starting the procedure for each tooth, the patient was asked to choose the envelope. Thus, the sequence of treatments was determined. The envelopes chosen for each treatment were discarded.

The teeth grouped in group R were treated with composite resin restoration without liner material, considered a control group.

The teeth grouped in group D received PBS CIMMO DTA® as indirect capping material of the cavity, followed by restoration of composite resin.

Sensitivity tests

Before starting the restorative treatment, dental sensitivity assessment was performed: Cold test: Using cotton in Cremer® balls, safe in clinical forceps (Duflex®), cooled with fluorethane gas, applied over the buccal surface of the tooth for 15s or until patient indicates painful sensation (Endo Ice® Spray, Maquira), for the Cold Test. The time from the beginning of the stimulus until its disappearance was counted (Time of Decline of pain). Percussion test: With the aid of the mouth mirror handle (Duflex®), the tooth was touched with light "taps", in the occlusal-apical and vestibule-lingual / vestibule-palate directions. Masticatory strength test: The patient performed masticatory movements under a bite device (Indusbello®, Londrina, PR, Brazil). The patient's perceptions of sensitivity were checked on a scale from 0 to 10 using the Visual Analogue Scale (VAS).

Restorative procedures

Pumice prophylaxis (SS White®, Rio de Janeiro, RJ, Brazil) and water were initially performed in order to remove residues and / or dental biofilm. Proceeding to the stage of topical anesthesia (Benzotop® 200mg, DFL, Jacarepaguá, RJ, Brazil), followed by local infiltrative anesthesia (Alphacaine® 2% DFL, Jacarepaguá, RJ, Brazil) and absolute isolation of the operative field.

It should be noted that the absolute isolation was performed prior to the cavity preparation, following the sanitary rules (Covid 19), to contain aerosols caused by the use of high speed.

The operative procedure was performed initially with spherical diamond tips (KG® Sorensen, Cotia, SP, Brazil) numbering compatible with the carious lesion (1011, 1012, 1013, 1014, 1016), until reaching the caries carefully, so as not to remove structure healthy dental. Then, carbide steel spherical drills, numbering compatible with the lesion, no. 2, 4 or 6 (KG Sorensen®, Cotia, SP, Brazil) were used at low speed (Contra-angle, Kavo®, Joinville, PR, Brazil) to remove carious tissue. Each diamond tip and Carbide drill was used a maximum of 4 times, after which they were discarded.

For restorations that needed to restore the shape of the proximal walls, wedges, preformed metal matrices and staples (Unimatrix®, TDV Pomerode-SC-Brasil) were used.

Subsequently, the cavities were restored, as described below:

In group R teeth, the following operative step was performed:

Conditioning with 37% phosphoric acid (Condac® 37, FGM, Joinville, SC, Brazil) was performed for 30 seconds on enamel and 15 seconds on dentin. Then the cavity was washed with the aid of a triple syringe using an air / water jet for 10 seconds.

The cavities received the restorative system composed of the Adper Single Bond2® adhesive, and the nano-particulate resin Filtek Z350XT® (3M ESPE Dental Products TM, St. Paul, MN, USA). The dentin substrate was left slightly moist, with the aid of cotton in Cremer® balls. Adhesive material was used, using a Cavibrush® microbrush brush, FGM, Joinville, SC, Brazil), strictly following the manufacturer's rules, used for this purpose; saturated for each covering, two consecutive layers of the enamel and dentin adhesive were applied, waited 30 seconds, continued with light air jets for 5 seconds and then the photoactivation was performed for 10 seconds with LED (Poly® Wireless , Kavo, Joinville-SC-Brazil), with a power of 600 ± 50 mW / cm².

The restorations were performed using the composite resin Filtek Z350 XT® (3M ESPE Dental Products TM, St. Paul, MN, USA) using the incremental oblique technique, in increments of a maximum of 2 mm in thickness, and each increment was photoactivated by 20 seconds, with LED (Poly® Wireless, Kavo, Joinville, SC, Brazil) final polymerization for 40s.

After the restorations were completed, absolute isolation was removed, then the sculpture was refined and occlusal adjustment was carried out, immediate finishing with thin diamond tips number 2135F, 3118F and 3195F (KG Sorensen®, Cotia, SP, Brazil), depending of the restored anatomical region. Polishing was carried out with abrasive silicone polishers for resins (Microdont®, Camanducaia, SP-Brazil) in medium (yellow) and superfine (white) granules and felt disc (Diamond®, FGM) with diamond paste (Diamond Excel® , FGM, Joinville, SC, Brazil).

In group D teeth, the same restorative step was also carried out, but prior to the acid conditioning step, PBS CIMMO DTA® cement was applied as a base for the dental cavity, following the manufacturer's instructions.

The PBS CIMMO DTA® Cement was handled in a sterile glass plate and spatula 24 (Duflex®), a portion of the cement powder and a drop of distilled water were dispensed (1: 1 ratio). Then, the manipulated material was inserted, with the aid of a dentin spoon (Duflex®), to the pulp wall of the cavity preparation. Using clinical forceps (Duflex®) and cotton in Cremer® balls, the cement was condensed at the bottom of the cavity, obtaining adaptation and removing excess moisture. Then, acid conditioning, adhesive application, restorative technique and polishing were performed as previously recommended for group R.

Clinical evaluations

The research participants had their personal records, anamnesis, as well as the type of treatment proposed inserted in a clinical form. However, only the operator, who performed the restorative procedures, had access to them. In another form, the values obtained in the Sensitivity Tests at 5 different moments were noted. The first tests, performed in the preoperative period and the others in the postoperative period. The evaluations were performed by a single examiner, trained by the researcher and not involved with the restorative procedures. The evaluations were noted on a specific form (Appendix B). The examiner was kept blind in all assessments.

It is noteworthy that: due to the health requirements imposed by the pandemic Covid 19, the evaluations were carried out by a single evaluator.

Sensitivity assessment

Sensitivity tests were performed before the restorative procedure, at 48 hours, 7, 15 and 30 days post-procedures. The analysis included: pain caused by thermal stimuli, percussion and bite.

For the thermal test, cotton was used in Cremer® balls, secured by clinical forceps (Duflex®), cooled with fluorethane gas (Endo Ice® Spray, Maquira) and applied over the buccal surface of the treated tooth, for 15s or even the patient indicates painful sensation. In the percussion test, with the aid of the mouth mirror handle (Duflex®), touches were made on the tooth with light "taps", in the occlusal-apical and vestibule-lingual / vestibule-palate directions. For the test of masticatory forces, the patient performed masticatory movements under a bite device (Indusbello®, Londrina, PR, Brazil).

The patients received a Visual Analogue Scale (VAS) (AMARAL and CALASANS, 2013) (Figure 1). Sensitivity perceptions were cataloged from 0 to 10. The scores determined were: 0 no pain, 1 to 2 mild pain, 3 to 5 moderate pain, 6 to 7 moderate pain slightly worse, 8 to 9 severe pain, 10 maximum pain .

The analyzes were tabulated in Microsoft exel and sent for statistical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years, with maximum age of 20 years.
* Periapical radiography for diagnosis with detection of the presence of carious lesion in premolar or permanent molar dentin.
* Lesion depth and cervical width of at least 1 mm, without pulp exposure.
* Presence of the antagonist, which must be a natural tooth, the same for adjacent teeth.
* Presence of vital pulp and absence of spontaneous painful symptoms.
* Presence of teeth without prior restorative treatment and oral health.

Exclusion Criteria:

* Patients who did not show up for post-operative evaluations.
* Patients who gave up participating in the study, after being included, for personal reasons.
* Patients tested positive for the SARS-Cov-2 virus, unable to be assessed for the required confinement.
* Treated patients in which the teeth presented, in the postoperative evaluations, the presence of inflammation and necrosis.

Ages: 18 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients from the Dental Office of the 14th GAC - Pouso Alegre (MG), Military Organization of the Brazilian Army. Therefore, all are male, as they belong to the military organization for men only.
Enrollment: 20 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative sensitivity in posterior teeth: before the procedure, 48 hours later, 7; 15 and 30 days later. Thermal test. | Sensitivity tests (thermal tests) were performed before the restorative procedure, 48 hours, 7, 15 and 30 days after the procedures
  Evaluate the postoperative sensitivity (thermal test) on posterior teeth, restored with CEMENT PBS CIMMO DTA®, as a lining material, and later restorations with composite resin.

SECONDARY OUTCOMES:
Evaluation of postoperative sensitivity in posterior teeth. Sensitivity test. Before the procedure, 48 hours later, 7; 15 and 30 days later. Percussion test. | Sensitivity tests (percussion tests) were performed before the restorative procedure, 48 hours, 7, 15 and 30 days after the procedures
  Evaluate the postoperative sensitivity (percussion test) on the posterior teeth, restored with CEMENT PBS CIMMO DTA®, as a covering material, and later restorations with composite resin.

OTHER OUTCOMES:
Evaluation of postoperative sensitivity in posterior teeth. Sensitivity test. Before the procedure, 48 hours later, 7; 15 and 30 days later. Masticatory strength test. | Sensitivity tests (masticatory strength tests) were performed before the restorative procedure, 48 hours, 7, 15 and 30 days after the procedures.
  Evaluate the postoperative sensitivity (masticatory forces test) on posterior teeth, restored with CEMENT PBS CIMMO DTA®, as a covering material, and later restorations with composite resin.

CONTACTS AND LOCATIONS:
Overall Officials: José Dias Silva Neto, Study Director — Universidade do Vale do Sapucaí
Locations (1):
- Univás, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It will be analyzed to the satisfaction